CLINICAL TRIAL: NCT04017169
Title: NO Reflow Phenomenon and Comparison to the Normal Flow Population Post Primary Percutaneous Coronary Intervention for ST Elevation Myocardial Infarction
Brief Title: No Reflow Phenomenon Incidence and Predictors
Acronym: NORM-PPCI
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: NORM PPCI
Record Dates: First submitted 2019-06-18; First posted 2019-07-12 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: No Reflow Phenomenon; STEMI
MeSH Terms: conditions — No-Reflow Phenomenon; ST Elevation Myocardial Infarction | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No reflow phenomenon: Those that during procedure experience no reflow phenomenon
  To define no reflow requires:
  • Angiographic evidence of reopening of occluded coronary artery and successful stent placement with no evidence of flow-limiting residual stenosis (<50%), dissection, vessel spasm, or thrombus burden
  and
  * Angiographic documentation of a TIMI flow grade ≤II, or
  * A TIMI flow grade III with a myocardial perfusion grade 0 or I, at least 10 min after the end of PCI procedure.
  Interventions: Other: No intervention as observational study
- No NRP: Normal angiographic coronary flow/blush post patent culprit vessel.
  Interventions: Other: No intervention as observational study

INTERVENTIONS:
Other: No intervention as observational study

SUMMARY:
Background No reflow phenomenon is described in up to 65% of patients undergoing primary percutaneous coronary intervention for ST elevation myocardial infarction (STEMI). It is known to be associated with worse outcomes but predictors of no reflow are not clearly described.

Objectives A single centre case-control observational study of patients presenting with acute myocardial infarction appropriate for PPCI comparing baseline clinical, biochemical and angiographic characteristics between patients with no reflow phenomenon and those without. Aiming to establish incidence for the UK population.

Secondary outcomes will be to gain further insight into those presenting with STEMI for PPCI and develop a risk model to guide management and clinical outcomes of patients to 30days.

Methods This study will prospectively recruit all consecutive patients attending a single centre for primary percutaneous coronary intervention for STEMI. Angiographic assessment of the recanalised epicardial vessel will be used to diagnose no reflow (reduced TIMI flow or blush grade). Baseline demographic, angiographic and biochemical characteristics and outcomes at 30days for reflow and no reflow cohorts will be statistically assessed and compared with logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presenting with ST elevation myocardial infarction
* Appropriate for Primary Percutaneous Coronary Intervention

Exclusion Criteria:

* Primary Percutaneous Coronary Intervention not performed eg due to non- flow- limiting coronary artery disease
* Unsuccessful PCI
* Thrombolysis
* Patients who do not survive the procedure to leave the catheterisation laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort is defined as all patients attending with ST elevation myocardial infarction undergoing primary percutaneous coronary intervention. Cases are those subjects who suffered no reflow phenomenon, with control comparators those that had TIMI III flow and grade III myocardial blush post procedure.
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of no reflow phenomenon | 0-2 days

SECONDARY OUTCOMES:
Predictors of no reflow phenomenon | 0-3 days
  Statistical analysis of multiple variables to find independent predictors
MACE outcomes | 30 days
  * Cardiovascular death
  * Death
  * Hearth Failure (Killip class III/IV)
  * MI
  * CVA
  * Repeat unplanned angiography
  * Repeat unplanned revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Rossington, BSc MBChB, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Castle Hill Hospital (Hull and east Yorkshire Hospitals NHS Trust), Cottingham, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No